CLINICAL TRIAL: NCT00499135
Title: Pharmacodynamic Study of Sunitinib Malate in Patients With Renal Cell Cancer and Other Advanced Solid Malignancies
Brief Title: Sunitinib Malate in Treating Patients With Unresectable or Metastatic Kidney Cancer or Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00245; NCI-2009-00245 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000552705; H-2007-0039; CO06902; CO 06902 (Other: University of Wisconsin Hospital and Clinics); 7898 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Adult Solid Neoplasm; Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — alovudine; Magnetic Resonance Spectroscopy; Sunitinib

ARMS (2):
- Schedule A (Experimental): Patients receive sunitinib malate PO QD in weeks 1-4. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Computed Tomography; Other: Fluorothymidine F-18; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Positron Emission Tomography; Drug: Sunitinib Malate
- Schedule B (Experimental): Patients receive sunitinib malate PO QD in weeks 1, 2, 4, and 5. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Computed Tomography; Other: Fluorothymidine F-18; Other: Pharmacological Study; Other: Positron Emission Tomography; Drug: Sunitinib Malate

INTERVENTIONS:
Other: Computed Tomography — Correlative studies
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Other: Fluorothymidine F-18 — Correlative studies
  Other Names: 18F-FLT; 3'-deoxy-3'-(18F) fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F 18
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Schedule A
Other: Pharmacological Study — Correlative studies
Other: Positron Emission Tomography — Correlative studies
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase I trial is studying the side effects and best way to give sunitinib malate in treating patients with unresectable or metastatic kidney cancer or other advanced solid tumors. Sunitinib malate may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the pharmacodynamic change using functional imaging (3'-deoxy-3'-[18F] fluorothymidine [FLT]-positron emission tomography [PET]/computed tomography [CT] scans) in patients with unresectable or metastatic clear cell renal cell carcinoma or other advanced solid malignancies treated with two different schedules of sunitinib malate.

II. Evaluate the objective response in patients treated with this drug.

SECONDARY OBJECTIVES:

I. Measure the change in plasma vascular endothelial growth factor (VEGF) levels and plasma hypoxia-inducible factor (HIF)1-alpha levels as a potential mechanism for vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI) failure and rapid tumor growth following VEGFR TKI withdrawal in these patients.

II. Correlate pharmacokinetics of this drug with response, unexpected toxicity, VEGF levels, HIF1-alpha levels, and FLT-PET/CT scan changes.

OUTLINE: Patients are assigned to 1 of 2 different treatment schedules of sunitinib malate.

SCHEDULE A: Patients receive sunitinib malate orally (PO) once daily (QD) in weeks 1-4. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

SCHEDULE B: Patients receive sunitinib malate PO QD in weeks 1, 2, 4, and 5. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell cancer; or other solid malignancy (excluding lymphoma) that is metastatic or unresectable and for which no standard curative therapy exists

  * For the renal cell cancer subset, a component of clear cell histology is required
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* Life expectancy > 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Serum calcium =< 12.0 mg/dL
* Total bilirubin normal
* Aspartate aminotransferase (AST) (serum glutamic oxalo-acetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times upper limit of normal (ULN), unless subjects have liver metastases, in which case both AST and ALT must be =< 5 x ULN
* Creatinine =< 2 times ULN OR creatinine clearance >= 40 mL/min for patients with creatinine levels above 2 x institutional normal
* All patients need to be willing to undergo planned pharmacodynamic assessments, including serial PET imaging, plasma markers, and pharmacokinetic sampling
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, experimental therapy or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (to grade < 1 or baseline) from clinically significant adverse events due to agents administered more than 4 weeks earlier (alopecia and fatigue excluded); clinical significance to be determined by investigator
* Patients may not be receiving any other investigational agents
* No prior treatment with an anti-VEGF agent allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* Patients with QTc prolongation (defined as a QTc interval greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities (per investigator discretion) are excluded
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mm Hg or higher or diastolic blood pressure of 90 mm Hg or higher) are ineligible
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within the past 28 days
  * Cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 12 months
  * History of pulmonary embolism within the past 12 months
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible; patients with a history of hypothyroidism are eligible provided they are currently euthyroid
* Patients with known brain metastases
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant or breastfeeding
* No concurrent therapeutic doses of coumarin-derivative anticoagulants, such as warfarin; Concurrent doses =< 2 mg/day allowed for prophylaxis of thrombosis, Concurrent low molecular weight heparin allowed provided prothrombin time (PT) international normalized ratio ( INR) =< 1.5
* No concurrent agents with proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide acetate)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05-22 (Actual); Primary Completion 2014-05-14 (Actual); Study Completion 2014-05-14 (Actual)

PRIMARY OUTCOMES:
Objective response | Up to 3 years
Plasma VEGF and HIF1-alpha levels | Up to 3 years
Standard uptake value as measured by 3'-deoxy-3'-[18F] fluorothymidine (FLT)-PET/CT scans | Up to 3 years

SECONDARY OUTCOMES:
Pharmacokinetic parameters (Cmax, Tmax, AUC, T1/2, and CL) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States